CLINICAL TRIAL: NCT05594914
Title: The Preliminary Efficacy and Safety of AK104 Plus Concurrent Chemoradiation Therapy in Unresectable Locally Advanced Esophageal Squamous Cell Carcinoma
Brief Title: AK104 Plus Concurrent Chemoradiation Therapy in Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of University of South China (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022KS-FL-13-02
Record Dates: First submitted 2022-10-15; First posted 2022-10-26 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK104 plus concurrent chemoradiation therapy (Experimental): AK104 10mg/kg plus TC regimen(paclitaxel liposome 135mg/m2, carboplatin AUC=5), once every 3 weeks (Q3W), induction treatment for 2 cycles; Subsequently, AK104 10 mg/kg plus TC regimen(paclitaxel liposome 135mg/m2, carboplatin AUC=5) is combined with radiotherapy(50Gy/25F) for 2 cycles.
  Interventions: Drug: AK104

INTERVENTIONS:
Drug: AK104 — AK104 plus TC regimen(paclitaxel liposome , carboplatin), once every 3 weeks (Q3W), induction treatment for 2 cycles; Subsequently, AK104 plus TC regimen is combined with radiotherapy for 2 cycles.

SUMMARY:
The purpose of this study is to assess the safety and efficacy of AK104 plus concurrent chemoradiation therapy in unresectable locally advanced esophageal squamous cell carcinoma

DETAILED DESCRIPTION:
AK104 10mg/kg plus TC regimen(paclitaxel liposome 135mg/m2, carboplatin AUC=5), once every 3 weeks (Q3W), induction treatment for 2 cycles; Subsequently, AK104 10 mg/kg plus TC regimen(paclitaxel liposome 135mg/m2, carboplatin AUC=5) is combined with radiotherapy(50Gy/25F) for 2 cycles. Assess disease efficiency( objective response rate; disease control rate; duration of overall response; time to resolve) and safety( adverse event).

ELIGIBILITY:
Inclusion Criteria:

* unresectable locally advanced esophageal squamous cell carcinoma; ECOG PS 0-1; At least one measurable lesion according to RESIST standard 1.1； not received anti-tumor treatment in the past

Exclusion Criteria:

* received immunotherapy in the past； Active hepatitis B, hepatitis C and other infectious diseases； Severe liver and kidney function, cardiovascular and cerebrovascular abnormalities

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
ORR | 24 months
  objective response rate
DCR | 24 months
  disease control rate
DoR | 24 months
  duration of overall response
TTR | 24 months
  time to resolve
AE | 24 months
  adverse event

SECONDARY OUTCOMES:
PFS | 24 months
  progression-free survival
OS | 24 months
  overall survival

IPD SHARING:
Plan to Share IPD: No